CLINICAL TRIAL: NCT06056310
Title: A Single Arm, Open Label, Phase 1b Study of Xevinapant in Combination With Weekly Cisplatin and Intensity-modulated Radiotherapy to Assess Safety and Tolerability in Participants With LA SCCHN, Suitable for Definitive Chemoradiotherapy (HyperlynX)
Brief Title: Phase 1b Safety Study of Xevinapant, Weekly Cisplatin, and RT in Participants With Unresected LA SCCHN (HyperlynX)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No major safety concerns were identified in HyperlynX study, but Lack of evidence of efficacy of meaningful clinical benefit.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS202359_0025; 2023-505796-76-00 (Other: EU CTIS)
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
Keywords: Unresected; Combination with CRT; Stage III; Stage IVA; Stage IVB; Oropharynx; Hypopharynx; Larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xevinapant + Cisplatin + IMRT (Experimental): Participants will receive xevinapant once daily from Day 1 to Day 14, per 3-week cycle (Each cycle is of 3 weeks). The first three cycles are given in combination with weekly cisplatin and radiotherapy, followed by 3 cycles of monotherapy xevinapant.
  Interventions: Drug: Xevinapant; Drug: Cisplatin; Radiation: intensity-modulated radiation therapy (IMRT)

INTERVENTIONS:
Drug: Xevinapant — Participants will receive xevinapant once daily from Day 1 to Day 14, per 3-week cycle (Each cycle is of 3 weeks). The first three cycles are given in combination with weekly cisplatin and radiotherapy, followed by 3 cycles of monotherapy xevinapant.
  Other Names: Debio 1143
Drug: Cisplatin — Participants will receive weekly cisplatin for 7 weeks on Cycle 1 Day 2 (C1D2), C1D9, C1D16, C2D2, C2D9, C2D16, and C3D2).
Radiation: intensity-modulated radiation therapy (IMRT) — Participants will receive 70 Gray (Gy) of IMRT in 35 fractions, 2 Gy/fraction, 5 days/week

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of Xevinapant when added to weekly cisplatin-based concurrent chemoradiotherapy (CRT) in the treatment of participants with unresectable locally advanced squamous cell carcinoma of the head and neck, suitable for definitive chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants having an Eastern Cooperative Oncology Group Performance Score (ECOG PS) of 0 - 1
* Histologically confirmed diagnosis in previously untreated Locally Advanced Squamous Cell Carcinoma of Head and neck (LA SCCHN) patient (Stage III, IVA, or IVB according to the American Joint Committee on Cancer [AJCC]/ Tumor Nodes and metastases (TNM) Staging System, 8th Edition) suitable for definitive Chemoradiotherapy (CRT), with one of the following primary sites: oropharynx (OPC) Human Papillomavirus (HPV)-negative, hypopharynx, and larynx
* Participant should be able to swallow liquids or has an adequately functioning feeding tube, gastrostomy, or jejunostomy in place. For participants requiring liquid nutrition at baseline or during the study including the follow-up period, access to liquid nutrition supply should be ensured
* Participant with evaluable tumor burden (measurable and/or non-measurable tumor lesions) assessed by CT scan and/or MRI, based on RECIST v 1.1.
* Adequate hematological, hepatic, and renal function as defined in the protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Primary tumor of nasopharyngeal, paranasal sinuses, nasal, or oral cavity, salivary, thyroid, or parathyroid gland pathologies, skin, or unknown primary site
* Metastatic disease (Stage IVC as per AJCC/TNM, 8th Edition)
* Existing need of a hearing aid or greater than or equal to (>=) 25 decibel shift over 2 contiguous frequencies on a pretreatment hearing test as clinically indicated
* Known history of infection with human immunodeficiency virus (HIV). If unknown history of HIV, an HIV screening test is to be performed and participants with positive serology for HIV-1/2 must be excluded
* Known gastrointestinal disorder with clinically established malabsorption syndrome and major gastrointestinal surgery in the last 12 months that may limit oral absorption
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (23):
- United States (5):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Karmanos Cancer Institute - PARENT, Detroit, Michigan
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
- Belgium (4):
  - Uza - Parent, Edegem
  - Universitair Ziekenhuis Gent - Medical Oncology, Ghent
  - Centre Hospitalier de l'Ardenne - PARENT, Libramont
  - Vitaz, Sint-Niklaas
- Hadassah University Hospital - Ein Kerem, Jerusalem, Israel
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam
  - Konkuk University Medical Center, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (4):
  - ICO Girona - Hospital Universitari de Girona Dr Josep Trueta - Servicio de Oncologia Medica, Girona
  - Clinica Universidad de Navarra (MAD) - Oncology Service, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz - Oncology, Madrid
  - Hospital Universitario Virgen del Rocio - Oncology Service, Seville
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202359_0025
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Participants received 3 cycles of oral solution of Xevinapant at a dose of 200 milligrams per day (mg/day) once daily from Day 1 to 14, per 3-week cycle. The first three cycles are given in combination with Cisplatin at dose of 40 milligrams per square meter (mg/m2) once daily on Cycle 1 Day 2 (C1D2, C1D9, C1D16, C2D2, C2D9, C2D16, and C3D2) With 70 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 35 fractions, 2 Gy/fraction, 5 days/week followed by 3 cycles of monotherapy of Xevinapant at a dose of 200 mg/day from Day 1 to 14, per 3-week cycle (Each cycle is of 3 weeks).
Period: Overall Study
Arm/Group | Sequence 1
Started | 18
Completed | 0
Not Completed | 18
Not completed — Other Reasons | 2
Not completed — Sponsor Request | 16

BASELINE CHARACTERISTICS:
Arm/Group | Sequence 1
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 1
  Ethnicity-Not Hispanic or Latino | 17
  Race-Asian | 11
  Race-Black or African American | 1
  Race-White | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)-Like Events
Description: DLT-like events defined as any of the following treatment-related adverse events (AEs) or lab abnormalities occurring during the 5-week DLT-like assessment period and assessed as related to the study intervention: Grade 4 asymptomatic neutropenia more than (>) 7 days; Grade 2-3 febrile neutropenia; Grade 4 thrombocytopenia without bleeding more than and equal to (>=) 5 days or Grade 2-3 with bleeding or requiring transfusion; Grade 2-3 nonhematologic toxicity (e.g., renal impairment based on eGFR, Grade 4 skin toxicity/mucositis interfering with treatment); less than (<) 60% planned cumulative dose of xevinapant or cisplatin due to AE; >2-week Radiation therapy (RT) delay due to AE; Grade >=2 ototoxicity worsening >=2 grades from baseline and considered treatment-limiting; Hy's Law DILI; Grade >=3 lab abnormalities; any life-threatening or Grade 5 toxicity.
Time Frame: Time from the first dose of study intervention day upto 35 days (5 weeks)
Population: DLT analysis set: all participants who received any study dose, met at least 1 of criteria: Had at least one DLT like event confirmed by SMC during DLT like assessment period or for whom ICE strategy led to DLT event, regardless of administered number of doses; Received at least 60% planned cumulative dose of xevinapant, cisplatin, regardless of completion in assessment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1
Number analyzed (Participants) | 18
Participants | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: AEs were defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. TEAEs were defined as AEs emerging or worsening after start of treatment until 30 days after end of treatment. Adverse events were coded according to the latest available version of the Medical Dictionary for Regulatory Activities (MedDRA). Treatment-Related TEAEs was defined as any AE considered as related to study treatment.
Time Frame: Screening up to end of treatment (Day 134) and then follow up every 3 months (assessed up to maximum 6 months)
Population: Safety analysis set (SAS) included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1
Number analyzed (Participants) | 18
Participants
  TEAEs | 18
  Treatment Related TEAEs | 18

3. Secondary Outcome: Absolute Estimated Glomerular Filtration Rate (eGFR) Values
Description: eGFR creatinine was evaluated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. Absolute values in eGFR was presented. Here, mL/min/1.73 m^2 is defined as milliliters per minute per 1.73 square meters.
Time Frame: At Cycle1 Day 4 (C1D4), C1D11, C1D18, C2D1, C2D4, C2D11, C2D18, C3D1, C3D4, C4D1, C5D1, C6D1 and End of treatment (Day 134) (each cycle is of 3 weeks)
Population: SAS included all participants who were administered any dose of any study intervention. Here" overall number of participants analyzed signified" participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Sequence 1
Number analyzed (Participants) | 17
mL/min/1.73 m^2
  C1D4 | 83.2080 (17.72417)
  C1D11: number analyzed (Participants) | 16
  C1D11 | 83.3678 (15.16465)
  C1D18: number analyzed (Participants) | 15
  C1D18 | 85.0461 (15.67478)
  C2D1: number analyzed (Participants) | 16
  C2D1 | 93.4136 (14.57590)
  C2D4: number analyzed (Participants) | 13
  C2D4 | 83.4911 (14.94634)
  C2D11: number analyzed (Participants) | 15
  C2D11 | 81.6135 (17.53286)
  C2D18: number analyzed (Participants) | 13
  C2D18 | 85.1155 (16.14240)
  C3D1: number analyzed (Participants) | 16
  C3D1 | 87.1169 (12.80356)
  C3D4: number analyzed (Participants) | 13
  C3D4 | 82.8900 (17.87483)
  C4D1: number analyzed (Participants) | 7
  C4D1 | 90.0343 (15.56475)
  C5D1: number analyzed (Participants) | 5
  C5D1 | 90.0000 (13.74773)
  C6D1: number analyzed (Participants) | 2
  C6D1 | 69.5000 (14.84924)
  End of treatment | 87.1937 (18.00761)

4. Secondary Outcome: Absolute Change From Baseline in eGFR
Description: eGFR creatinine was evaluated using CKD-EPI formula. Absolute change from baseline in eGFR was presented.
Time Frame: Baseline, C1D4, C1D11, C1D18, C2D1, C2D4, C2D11, C2D18, C3D1, C3D4, C4D1, C5D1, C6D1 and End of treatment (Day 134) (each cycle is of 3 weeks)
Population: SAS included all participants who were administered any dose of any study intervention. Here "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Sequence 1
Number analyzed (Participants) | 18
mL/min/1.73 m^2
  Baseline | 89.6908 (13.35296)
  C1D4: number analyzed (Participants) | 17
  C1D4 | -7.1908 (10.69578)
  C1D11: number analyzed (Participants) | 16
  C1D11 | -8.2532 (17.46117)
  C1D18: number analyzed (Participants) | 15
  C1D18 | -5.8696 (6.03911)
  C2D1: number analyzed (Participants) | 16
  C2D1 | 2.3052 (10.00664)
  C2D4: number analyzed (Participants) | 13
  C2D4 | -6.3632 (13.50060)
  C2D11: number analyzed (Participants) | 15
  C2D11 | -9.3021 (16.44543)
  C2D18: number analyzed (Participants) | 13
  C2D18 | -4.7388 (12.75881)
  C3D1: number analyzed (Participants) | 16
  C3D1 | -2.9103 (14.80991)
  C3D4: number analyzed (Participants) | 13
  C3D4 | -6.7050 (14.90582)
  C4D1: number analyzed (Participants) | 7
  C4D1 | -3.3451 (25.03351)
  C5D1: number analyzed (Participants) | 5
  C5D1 | -5.3312 (12.52264)
  C6D1: number analyzed (Participants) | 2
  C6D1 | -26.5000 (7.77817)
  End of treatment: number analyzed (Participants) | 17
  End of treatment | -2.4789 (16.82505)

5. Secondary Outcome: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 Criteria as Assessed by Investigator
Description: OR is defined as the number of participants who have a best overall response of complete response (CR) or partial response (PR) CR: Disappearance of target and non-target lesions and normalization of tumor markers.
  PR: At least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Non target lesions must be non-progressive disease.
Time Frame: Up to approximately 6 months
Population: FAS included all participants who were administered any dose of any study intervention. As pre-specified in statistical analysis plan (SAP), efficacy analysis was not conducted in this study (samples were not processed) and therefore data could not be analyzed and reported in this outcome measure.
Groups:
- Sequence 1: Participants received 3 cycles of oral solution of Xevinapant at adose of 200 milligrams per day (mg/day) once daily from Day 1 to14, per 3-week cycle. The first three cycles are given in combinationwith Cisplatin at dose of 40 milligrams per square meter (mg/m2)once daily on Cycle 1 Day 2 (C1D2, C1D9, C1D16, C2D2, C2D9, C2D16,and C3D2) With 70 Gray (Gy) of intensity modulated radiationtherapy (IMRT) in 35 fractions, 2 Gy/fraction, 5 days/week followedby 3 cycles of monotherapy of Xevinapant at a dose of 200 mg/dayfrom Day 1 to 14, per 3-week cycle (Each cycle is of 3 weeks).
Arm/Group | Sequence 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression Free Survival (PFS) According to RECIST Version 1.1 Criteria as Assessed by Investigator
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on Blinded Independent Central Review (BICR), or death due to any cause, whichever occurs first. According to RECIST 1.1, progressive disease (PD) was defined as a 20% relative increase in the sum of diameters (SOD) of target lesions, taking as reference the nadir SOD and an absolute increase of >5 millimeter (mm) in the SOD, or the appearance of new lesions.
Time Frame: Time from randomization to the first documented disease progression, or death due to any cause, whichever occurs first (up to approximately 6 months)
Population: Full Analysis Set included all participants who were randomized to study treatment. As pre-specified in SAP, efficacy analysis was not conducted in this study (samples were not processed) and therefore data could not be analyzed and reported in this outcome measure.
Arm/Group | Sequence 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Locoregional Control (LRC) According to RECIST Version 1.1 Criteria As Assessed by Investigator
Description: LRC is defined as the time from date of the first treatment until date of the first occurrence of progression at the site of the primary tumor or the locoregional lymph nodes.
Time Frame: Time from date of the first treatment until date of the first occurrence of progression at the site of the primary tumor or the locoregional lymph nodes or End of Study, assessed approximately up to 6 months
Population: as for outcome 6
Arm/Group | Sequence 1
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to Subsequent Systemic Cancer Treatments
Description: Time to subsequent systematic cancer treatments was defined as time from date of the first treatment administration until the start date of the first subsequent systemic cancer treatment for squamous cell carcinoma of the head and neck (SCCHN).
Time Frame: Time from date of the first treatment administration until the start date of the first subsequent systemic cancer treatment for SCCHN or End of study, assessed up to approximately 6 months
Population: as for outcome 6
Arm/Group | Sequence 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Screening up to end of treatment (Day 134) and then follow up every 3 months (assessed up to maximum 6 months)
Arm/Group | Sequence 1
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1 (N=18)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1 (N=18)
Anaemia (Blood and lymphatic system disorders) | 5 (7)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Central serous chorioretinopathy (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Localised oedema (General disorders) | 1 (2)
Mucosal inflammation (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (3)
Candida infection (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tongue fungal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (6)
Amylase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Lipase increased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (4)
Weight decreased (Investigations) | 6 (6)
White blood cell count decreased (Investigations) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypogeusia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (3)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT06056310/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT06056310/SAP_001.pdf